CLINICAL TRIAL: NCT06505746
Title: Adelphi Real World Metastatic Urothelial Cancer Disease Specific Programme: Study of Real-world Data to Evaluate Patient Characteristics, Treatment Pattern and Healthcare Resource Utilisation of Locally Advanced or Metastatic Urothelial Cancer (La/mUC) at First-line Setting Post Avelumab Reimbursement in South Korea and Saudi Arabia
Brief Title: A Study of Real-world Treatment of Adults With Urothelial Cancer in South Korea and Saudi Arabia
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 7465-MA-3515
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Bladder cancer; LA/mUC
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LA/mUC patients: LA/mUC patient record-based survey of medical oncologists and urologists in Saudi Arabia and South Korea.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No investigational drug will be administered to participants in this study.

SUMMARY:
Cancer in the bladder lining (urothelial cancer) can be treated in many ways. One way is to directly attack cancer cells. Enfortumab vedotin is a treatment that can do this. Another way is to help the body's immune system find and attack cancer cells. Avelumab is a treatment that can do this. Both treatments were recently approved in some countries.

Doctors have standard clinical practice guidelines to help them treat people with cancer. This study is about collecting information on how adults with urothelial cancer are treated in standard clinical practice. The people in this study will have locally advanced or metastatic urothelial cancer. Locally advanced means the cancer has spread to tissue close by.

Metastatic means the cancer has spread to other parts of the body.

The goal of this study is to learn how people with urothelial cancer receive medical care in clinics in South Korea and Saudi Arabia. The main goals are to learn more about the people receiving treatments, and the treatments they receive.

This study is about collecting information only. The individual's doctor decides on treatment, not the study sponsor (Astellas).

Information will be collected from the people's medical records. This will include 12 months before treatment starts, and during treatment. Also, doctors will answer questions in interviews and surveys about how they care for people with urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

Physician sample:

* Medical oncologist or urologist (Medical oncologists only in Saudi Arabia. A minimum of 15 medical oncologists in South Korea, increased where possible, with the remaining sample consisting of urologists)
* Personally responsible for treatment and management of LA/mUC patients
* At least 50 percent of time spent in management of patients
* See a minimum of 4 LA/mUC patients per month
* Accept all survey rules and requirements

Patient sample:

* Confirmed/physician assessed diagnosis of LA/mUC
* Patient is not currently enrolled in a clinical trial

Exclusion Criteria:

* Patients currently enrolled in a clinical trial
* Patients participating in, or who have previously participated, in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: LA/mUC patients being treated by medical oncologists and urologists in Saudi Arabia and South Korea. Patients will be sampled within a routine care setting in that they are consulting a physician through a pre-planned appointment.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Demographics associated with LA/mUC patients at various stages of treatment pathway | Day 1
  Demographics of interest will be recorded.
Clinical characteristics associated with LA/mUC patients at various stages of treatment pathway | Day 1
  Clinical characteristics of interest will be recorded.
Therapies received at data collection and any therapies previously received for LA/mUC. | Day 1
  Details of current and previous therapies received for LA/mUC will be recorded.

SECONDARY OUTCOMES:
Healthcare resource utilization of 1L and 2L+ LA/mUC patients | Day 1
  LA/mUC Healthcare resources will be recorded.
Current molecular/genetic testing patterns in LA/mUC patients | Day 1
  Tumor biomarker, genetic tests results and PD1/PD-L1 expression status will be recorded.
Current diagnostic tools in LA/mUC patients | Day 1
  Tests and assessments used to diagnosis patient's LA/mUC will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Singapore Pte. Ltd.
Locations (1):
- KR00001, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.